CLINICAL TRIAL: NCT01102036
Title: Effects of Cultura Yoghurt in Relation to Transit Time and Digestive Discomfort During 2 Weeks of Treatment in Comparison to Placebo in Healthy Women and Men
Brief Title: Effects of Cultura Yoghurt in Relation to Transit Time and Digestive Discomfort in Healthy Women and Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Good Food Practice, Sweden (Industry)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Birgitta Sundberg, Director clinical trials, Good Food Practice, Sweden
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C-X-Ray U-09-017
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2010-04

CONDITIONS: Constipation
Keywords: Transit time; constipation; gut regularity; defecation frequency; Colonic transit time
MeSH Terms: conditions — Constipation | interventions — Yogurt; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoghurt without probiotics (Placebo Comparator): Yoghurt without probiotic bacteria
  Interventions: Other: Yoghurt without probiotics
- Cultura yoghurt (Active Comparator): Cultura yoghurt with L casei F19, acidophilus La5 adn B lactis Bb 12
  Interventions: Other: Cultura L casei F19, acidophilus La5 , B lactis Bb 12

INTERVENTIONS:
Other: Cultura L casei F19, acidophilus La5 , B lactis Bb 12 — 2 weeks consumption,250 ml/day
  Other Names: Cultura probiotic yoghurt; Yoghurt without prbiotics
  Arms: Cultura yoghurt
Other: Yoghurt without probiotics — Yoghurt without probiotics
  Arms: Yoghurt without probiotics

SUMMARY:
The aim of this study is to determine the effect of cultura yoghurt on transit time and digestive discomfort during 2 weeks of treatment in comparison to placebo in healthy women and men.

DETAILED DESCRIPTION:
Transit time is the time it takes for a substance to pass through the gut. The major part of the transit is spent in the large bowel is therefore mainly a colonic event. It has been observed that slow transit time is associated with high prevalence of large bowel disorders. The objectives of this study is to:

* determine the effect on mean transit time after 2 weeks intake of a investigational products using radio-opaque sulphate impregnated polyethylene pellets as markers.
* determine effect of investigational products on total symptom score according to Bristol Stool Form (BSF)
* determine effect of investigational products in gastrointestinal symptoms
* determine safety of intake of the investigational products

ELIGIBILITY:
Inclusion Criteria:

* Female and Males
* Healthy
* BMI 19-29 at visit 1
* Age 18 and 60 years at visit 1
* Defecation 3-4 times per week or every second to third day (Bristol Stool Form) during the run-in
* Transit time 35 and 72 hours calculated from the abdominal X-ray at visit 3
* Signed written informed consent

Exclusion Criteria:

* Use of probiotics food or supplements during the study
* Past history of digestive disease
* Previous complicated GI surgery
* Oral use of antimicrobial medication or antimicrobial prophylaxis 4 weeks prior to screening visit
* Use of laxatives (medication or dietary supplements) during the study.
* Pregnant or lactating or wish to become pregnant during the period of the study
* Lack of suitability for participation in the trial, for any reason, as judged by the personnel at KPL Good Food Practice AB

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in transit time between treatments | February 2010-June 2010
  To determine the effect on mean transit time after 2 weeks intake of investigational products using radio-opaque barium sulphate impregnated polyethylen capsules. These capsules will be consumed during 3 days and thereafter an x-ray image will be taken over the bowel. The capsulese will then be calculated to determine the colonic transit time

SECONDARY OUTCOMES:
Change between treatments on Bristol Stool Form (BSF)symptoms scores | February 2010-June2010
  To determine the effect of Cultura yoghurt on the total symptom score according to Bristol Stool Form (BSF) scale during 2 weeks of treatment in comparison to placebo in healthy women and men
Change between treatments on gastrointestinal symptoms according to Bristol Stool Form | February 2010-June 2010
  To determine the effect of Cultura yoghurt on gastrointestinal symptoms according to the Bristol Stool Form (BSF) after 2 weeks treatment of investigational products

CONTACTS AND LOCATIONS:
Overall Officials: Lars Magnusson, CEO, Study Director — Good Food Practice, Uppsala, Sweden
Locations (1):
- Good Food Practice, Uppsala, Sweden